CLINICAL TRIAL: NCT05417633
Title: RayOne EMV Mini-monovision - Efficiency and Safety of 3 Grades of Mini-monovision
Acronym: EMV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Somich, s.r.o. (Other)
Responsible Party: Principal Investigator, Tomas Benda, MD, FEBO, head of the department, Somich, s.r.o.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Somich
Record Dates: First submitted 2022-05-02; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Cataract Senile; Presbyopia
Keywords: Intraocular lens enhanced; minimonovision
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): monovision 0.25 - 0.74 D
  Interventions: Procedure: intraocular lens - RayOne EMV (Rayner Surgical GmbH,Berlin, Deutschland)
- Group 2 (Active Comparator): monovision 0.75 -1.24 D
  Interventions: Procedure: intraocular lens - RayOne EMV (Rayner Surgical GmbH,Berlin, Deutschland)
- Group 3 (Active Comparator): monovision 1.24 - 1.75
  Interventions: Procedure: intraocular lens - RayOne EMV (Rayner Surgical GmbH,Berlin, Deutschland)

INTERVENTIONS:
Procedure: intraocular lens - RayOne EMV (Rayner Surgical GmbH,Berlin, Deutschland) — Inducing different values of monovision

SUMMARY:
Aim:To determine the effectiveness and subjective satisfaction of patients with bilateral cataract surgery and implantation of intraocular lens (IOL) RayOne EMV with enhanced optic, using different degrees of mini-monovision (up to 0.74, between 0.75 -1.24 and 1.25-1.75). To compare individual groups between themselves . In particular, we would like to compare the independence of spectacle correction when looking into the distance, at medium distance and at reading distance.

DETAILED DESCRIPTION:
Purpose: To determine the effectiveness and subjective satisfaction of patients with bilateral cataract surgery and implantation of intraocular lens (IOL) RayOne EMV with enhanced optic, using different degrees of mini-monovision (up to 0.74, between 0.75 -1.24 and 1.25-1.75). To compare individual groups between themselve

Preoperative examination - Eye dominance - hole in card method Argos optical biometrics (Movu, Inc., CA, U.S.) Barrett's formulas (Barrett universal II) will be used to calculate the optimal IOL. A RayOne EMV lens with a planned postoperative spherical equivalent (SE) of -0.25 to 0.25 will be implanted in the dominant eye. A lens with a planned SE of -0.25 to -0.74 will be implanted in the non-dominant eye in the first group, -0.75 to -1.24 in the second group and -1.25 to -1.75 in the third group.

Surgery Standard course of surgery, corneal incision at No. 12, combination of topical and intracameral anesthesia, implantation of IOL into the capsular bag, primary posterior capsulorhexis (PPCCC) performed after implantation.

Postoperative evaluation In addition to standard postoperative examinations (anterior segment condition, intraocular pressure), the resulting refraction will be monitored postoperatively (3 and 6 months after second eye surgery) using an autorefractometer.

Uncorrected (UCVA) and corrected distance visual acuity (DCVA) will be examined using projection optotypes. Uncorrected (UIVA) medium distance visual acuity (60 cm) and uncorrected (UNVA) and corrected (CNVA) near visual acuity (30 cm) using standardized EDTRS reading tables. All values of visual acuity will be examined monocularly and binocularly (bUCVA, bDCVA, bUNVA, bCNVA, bUIVA). Visual acuity values will be expressed in logMAR.

Binocular Contrast sensitivity will be examined using a Glaretester CGT 1000 instrument (Takagi, Seiko Co. Ltd., Nagano, Japan) at a distance (test distance) of 30 cm, 60 cm 5 m. (day), type of glare, low glare, presentation duration of test target 0.8 s, presentation interval of test target 2 s. The resulting values will be expressed numerically and graphically in comparison with the standard .

Patients will be asked to complete questionnaires:

1. the occurrence of secondary visual symptoms (eg halo - ring around the light source, glare - fog around the light source and starbursts - rays around the light source). Patients will rate these side effects on a scale of 0 - 5 (0 - none, 1 - very mild, 2 - mild 3 - moderate 4 - severe 5 - very severe).
2. for independence on glasses a) at close range b) at medium distance c) at a distance. Patients rate on a scale of 1 - 5 (1 - never uses glasses, 2 - exceptionally uses glasses 3 - occasionally uses glasses 4 - often uses glasses 5 - always uses glasses).
3. Satisfaction with the result of the operation. Patients rate on a scale of 1 - 5 (1 - very satisfied 2 - rather satisfied 3 - neutral 4 - rather dissatisfied 5 - very dissatisfied).

6. Statistical analysis - descriptive data describing the group of patients and visual, refractive results and contrast sensitivity and questionnaires will be processed. The Wilcoxon signed-rank test will be used to compare preoperative and postoperative visual acuity. The Mann-Whitney U test will be used to compare visual symptoms and patient satisfaction in each group

ELIGIBILITY:
Inclusion Criteria:

- bilateral senile cataract

Exclusion Criteria:

* corneal astigmatism greater than 0.75 diopters (D)
* difference in the planned dioptric value of intraocular lens (IOL) over 2 D (calculated for bilateral emetropia)
* perioperative complications not allowing proper implantation and centering of IOL in the lens bag
* time between surgeries of both eyes greater than 1 month
* eye disease, which could reduce visual acuity
* previous refractive surgeries
* systemic diseases that could affect postoperative visual acuity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-21 (Estimated)

PRIMARY OUTCOMES:
visual acuity (VA) | 3-6 months
  uncorrected for distance (UDVA), intermediate distance (UIVA), near (UNVA) corrected for distance (CDVA), intermediate distance (CIVA), near (CNVA)
sS Subjective satisfaction | 3-6 months
  questionnaire of subjective satisfaction, dependence on glasses, incidence of secondary visual phenomena - scale 1-5

SECONDARY OUTCOMES:
contrast sensitivity | 3-6 months
  Glaretester

CONTACTS AND LOCATIONS:
Overall Officials: Eliska Studena, MSc, Study Director — Somich, s.r.o.
Locations (1):
- Somich, Karlovy Vary, Czechia

IPD SHARING:
Plan to Share IPD: No
one researcher

REFERENCES:
- [Background] Boerner CF, Thrasher BH. Results of monovision correction in bilateral pseudophakes. J Am Intraocul Implant Soc. 1984 Winter;10(1):49-50. doi: 10.1016/s0146-2776(84)80077-4. PMID 6706816
- [Background] Rodov L, Reitblat O, Levy A, Assia EI, Kleinmann G. Visual Outcomes and Patient Satisfaction for Trifocal, Extended Depth of Focus and Monofocal Intraocular Lenses. J Refract Surg. 2019 Jul 1;35(7):434-440. doi: 10.3928/1081597X-20190618-01. PMID 31298723
- [Background] Shen Z, Lin Y, Zhu Y, Liu X, Yan J, Yao K. Clinical comparison of patient outcomes following implantation of trifocal or bifocal intraocular lenses: a systematic review and meta-analysis. Sci Rep. 2017 Mar 28;7:45337. doi: 10.1038/srep45337. PMID 28422087
- [Background] Abdelrazek Hafez T, Helaly HA. Spectacle Independence And Patient Satisfaction With Pseudophakic Mini-Monovision Using Aberration-Free Intraocular Lens. Clin Ophthalmol. 2019 Oct 31;13:2111-2117. doi: 10.2147/OPTH.S215229. eCollection 2019. PMID 31802840
- [Background] Wilkins MR, Allan BD, Rubin GS, Findl O, Hollick EJ, Bunce C, Xing W; Moorfields IOL Study Group. Randomized trial of multifocal intraocular lenses versus monovision after bilateral cataract surgery. Ophthalmology. 2013 Dec;120(12):2449-2455.e1. doi: 10.1016/j.ophtha.2013.07.048. Epub 2013 Sep 23. PMID 24070808
- [Background] de Vries NE, Nuijts RM. Multifocal intraocular lenses in cataract surgery: literature review of benefits and side effects. J Cataract Refract Surg. 2013 Feb;39(2):268-78. doi: 10.1016/j.jcrs.2012.12.002. PMID 23332253
- [Result] Greenstein S, Pineda R 2nd. The Quest for Spectacle Independence: A Comparison of Multifocal Intraocular Lens Implants and Pseudophakic Monovision for Patients with Presbyopia. Semin Ophthalmol. 2017;32(1):111-115. doi: 10.1080/08820538.2016.1228400. Epub 2016 Oct 28. PMID 27792408